CLINICAL TRIAL: NCT02659566
Title: Impact of Antimalarial Treatment on Measures of T Cell Suppression/Regulation in Healthy Adults From Ouelessebougou, Mali
Brief Title: Impact of Antimalarial Treatment on Measures of T Cell Suppression/Regulation in Healthy Adults From Doneguebougou, Mali
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999916051; 16-I-N051
Record Dates: First submitted 2016-01-15; First posted 2016-01-20 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06-12

CONDITIONS: Malaria
Keywords: Markers; Parasitemia; Coartem; Plasmodium; Infection
MeSH Terms: conditions — Malaria; Parasitemia; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

Malaria is a disease that affects many people in the country of Mali and other parts of Africa. It is caused by germs that are spread by mosquito bites. Malaria may be mild, but can also be serious or can lead to death if not diagnosed and treated promptly. Children younger than 5 years and pregnant women are at highest risk of malaria. Researchers want to better understand how malaria infection suppresses the immune system. They want to compare a group of adults who receive antimalarial treatment to a group that does not receive it.

Objective:

To investigate the effect of antimalarial treatment at the beginning of the dry season on the immune system and malaria episodes.

Eligibility:

Healthy adults ages 18-60 who live in the area of Doneguebougou, Mali.

Design:

Participants will be screened with a physical exam and health questions.

If participants are found to be sick at the screening visit, they will get initial care at the study clinic free of charge. They may get referrals for consultation.

Participants will be randomly assigned to a group. One group will get an approved antimalarial drug called Coartem . The other will not receive it.

Participants in the Coartem group will take the drug for 3 days.

All participants will have blood tests.

Al participants will be seen about once a month for about 1 year. At each visit, they will be asked how they are feeling and be examined. Blood will be drawn.

If participants become sick at any time, they will come to the clinic to be examined.

DETAILED DESCRIPTION:
Malaria, caused by Plasmodium falciparum, is a devastating disease that causes significant mortality and morbidity both directly and indirectly in endemic regions. Lower all-cause mortality in children under five years of age have resulted from better malaria transmission control measures in endemic regions.

It has been seen in multiple studies that malaria infection, including asymptomatic carriage, suppresses or modulates the immune system; how exactly this suppression is achieved is unclear. Currently, efforts to develop long-lasting, effective vaccines to combat malaria have not been successful. One of the impediments of concern is poor immune response to the vaccine candidates. Understanding the immunomodulatory effects of malaria infection to vaccine responses and to subsequent malaria infection is thus key in these efforts.

In order to further understand how the presence of parasitemia may modulate the immune system, we propose to study the effects of treating a portion of adult volunteers with a treatment course of artemether/lumefantrine (Coartem ) at the beginning of the dry season (approximately January) in Ouelessebougou, Mali to clear parasitemia carriage during the dry season and following them for the next 10-12 months through an entire dry and wet season. We will enroll 50% blood smear or polymerase chain reaction (PCR) positive volunteers and distribute them equally into two groups at the beginning of the dry season, those who receive or do not receive antimalarial treatment. These subjects will then be followed monthly throughout the dry and rainy seasons to determine the effect of this treatment on T cell markers of suppression/regulation and the incidence of asymptomatic malaria infection and clinical malaria. We hypothesize that markers of T cell suppression/regulation throughout the dry season will be lower in adults who receive a single pre-emptive treatment with Coartem .

ELIGIBILITY:
* INCLUSION CRITERIA:

A study participant must satisfy the following criteria to be enrolled in this study:

* Provide individual informed consent
* Adult between ages of 18 and 60
* Willingness to have blood samples stored for future research
* Known resident of Ouelessebougou or surrounding area

EXCLUSION CRITERIA:

A subject will be excluded from participating in this trial if any one of the following criteria is fulfilled:

* Known to be pregnant (by history) or positive pregnancy test
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, hematological, oncologic, psychiatric, or renal disease by history and/or physical examination that may impact the subject s overall health and immune system
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and comply with the study protocol
* Use of chronic (greater than or equal to14 days) oral or intravenous corticosteroids (excluding topical or nasal) at immunosuppressive doses (i.e., prednisone >10 mg/day) or immunosuppressive drugs within 30 days of Study Day 0
* Receipt of Coartem within less than 14 days from Study Day 0
* Known allergies or contraindications (such as significant cardiac disease prolonged QTc >450 ms; currently taking medications that may prolong your QTc; serious side effects from Coartem in the past) to study treatment (Coartem [artemether/lumefantrine])
* Receipt of investigational malaria vaccine within the last 5 years
* Enrollment in another investigational trial during the study period (participating in screening for other investigational trials is permitted)
* Tested positive for HIV or Hepatitis B or Hepatitis C.
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a participant participating in the trial, interfere with the evaluation of the study objectives, or would render the subject unable to comply with the protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 290 (Actual)
Dates: Start 2016-01-15; Primary Completion 2018-06-12 (Actual); Study Completion 2018-06-12 (Actual)

PRIMARY OUTCOMES:
To measure the percentage of T cells expressing PD-1 during scheduled visits by comparing markers of T cell suppression/regulation in adults (specifically PD-1) who receive or do not receive antimalarial treatment at the beginning of dry season ... | Twelve months

CONTACTS AND LOCATIONS:
Overall Officials: Michal Fried, Ph.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Ouelessebougou Clinical Research Center, Bamako, Mali

REFERENCES:
- [Background] Cunnington AJ, Riley EM. Suppression of vaccine responses by malaria: insignificant or overlooked? Expert Rev Vaccines. 2010 Apr;9(4):409-29. doi: 10.1586/erv.10.16. PMID 20370551
- [Background] Illingworth J, Butler NS, Roetynck S, Mwacharo J, Pierce SK, Bejon P, Crompton PD, Marsh K, Ndungu FM. Chronic exposure to Plasmodium falciparum is associated with phenotypic evidence of B and T cell exhaustion. J Immunol. 2013 Feb 1;190(3):1038-47. doi: 10.4049/jimmunol.1202438. Epub 2012 Dec 21. PMID 23264654
- [Background] Moormann AM, Snider CJ, Chelimo K. The company malaria keeps: how co-infection with Epstein-Barr virus leads to endemic Burkitt lymphoma. Curr Opin Infect Dis. 2011 Oct;24(5):435-41. doi: 10.1097/QCO.0b013e328349ac4f. PMID 21885920